CLINICAL TRIAL: NCT06258213
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Doses Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral ABP-745 Administration in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral ABP-745 Administration in Healthy Volunteers
Acronym: ABP-745
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: ABP-745-101
Record Dates: First submitted 2024-01-29; First posted 2024-02-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Gout; Acute Gout Flare; Gout Flares
Keywords: acute gout flare; gout flares; tophi; chronic pain
MeSH Terms: conditions — Gout; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- ABP-745 (Active Comparator)
  Interventions: Drug: ABP-745

INTERVENTIONS:
Drug: ABP-745 — 0.5, 5 or 25 mg tablet
  Arms: ABP-745
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, dose-escalation study will be conducted in healthy volunteers. This study will evaluate the safety, tolerability, and pharmacokinetics (PK) of ABP-745 following single (Part 1) and multiple (Part 2) oral doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers, aged 18 and 55 years (inclusive) at the time of signing the informed consent form (ICF).
* Body mass index (BMI) range within 18 ~ 30 kg/m2 (inclusive), and body weight of ≥ 50.0 kg for male and ≥ 45.0 kg for female.
* Generally healthy based on medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory tests.
* Female volunteers of child-bearing potential must agree to use effective contraceptive methods from the screening period to 90 days after the last dose of the investigational product (IP).

Exclusion Criteria:

* Difficulties in venous blood collection or history of dizziness when encountering blood or needles.
* Has received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month or 5 times half-life (whichever is longer) prior to the first dose of IP.
* Has a history of gastrointestinal (such as duodenal ulcer, alimentary tract hemorrhage, gastro esophageal reflux disease (GERD), etc.), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs as determined by the Investigator (or Sub-investigator).
* Has the medical history (including past and present) of other significant diseases (including but not limited to pulmonary, cardiovascular, gastrointestinal, hematological, endocrinological and metabolic disease, immunological, dermatological, malignant diseases, mental and nervous systems, and other related diseases) or any other disease/ailment at the discretion of the Investigator (or Sub-investigator).
* Any medication (prescription and nonprescription) within 14 days or 5 times the half-life (whichever is longer) prior to the first dose of IP. (Excluding oral contraceptives, or topical ointments at the discretion of the Investigator (or Sub-investigator)).
* A known history of drug abuse within 2 years before the screening; or positive drug abuse test at screening.
* Blood donation or blood loss of more than 400 mL within 3 months before the screening.
* Smoking history (≥ 5 cigarettes per day) within 3 months before the screening, or cannot abstain from any tobacco products during the study.
* Positive screening test for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV) antibody.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (Safety and Tolerability) | Up to Day 14

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters including peak plasma concentration (Cmax) | Up to Day 11
Urine pharmacokinetic parameters including amount excreted in urine over the sampling interval (Ae) | Up to Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No